CLINICAL TRIAL: NCT05681533
Title: Tissu Adipeux épicardique et rigidité artérielle Chez Les Personnes Vivant Avec un diabète
Brief Title: Epicardial Adipose Tissue and Arterial Stiffness in People Living With Diabetes (METAB-CV-PWV)
Acronym: METAB-CV-PWV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220876
Record Dates: First submitted 2022-12-07; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-11

CONDITIONS: Diabetic Patients
Keywords: Diabet; arterial stiffness; pericardial adipose tissue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: CT scan — coronary calcium score measurement by CT scan

SUMMARY:
The present study is a retrospective and prospective current care cohort that will allow us to evaluate the relationship between epicardial fat volume and increased arterial stiffness in a person living with diabetes.

DETAILED DESCRIPTION:
Epicardial adipose tissue is considered as the cardiac visceral fat and is associated with increased cardiovascular risk, for example in diabetes. Thus, the mechanisms involved seem to be related to myocardial lipotoxicity; atherosclerosis in connection with inflammation and secretion of proinflammatory factors such as cytokines but also insulin resistance.

In this context, the investigators hypothesize that epicardiac adipose tissue volume will be higher in patients with increased arterial stiffness than in those without. In this study, the investigators will then try to verify the existence of a relationship between pericardial adipose tissue volume and increased arterial stiffness in people living with diabetes.

To do this, the investigators will analyze the results of measurements of pericardial fat volume, coronary calcium score, and pulse wave velocity in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for participation in the study if:

* They are informed and have not objected to participating in the research.
* They have type 1 or 2 diabetes.
* They perform a coronary calcium score measurement by CT scan and a pulse wave velocity assessment during their routine care practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 1 or 2 diabetic patients who perform coronary calcium score measurement by CT scan and pulse wave velocity assessment as part of their routine care practice.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Epicardial fat volume | the inclusion visit
  Epicardial fat volume will be determined using cardiac CT scan without contrast injection.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel COSSON, Pr, Principal Investigator — APHP, Hospital Avicenne
Locations (1):
- endocrinologie site, Avicenne hospital, Bobigny, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koutcha ON, Tatulashvili S, Sritharan N, Boutouyrie P, Rezgani I, Boubaya M, Mariko ML, Allard L, Sal M, Bloch-Queyrat C, Zerguine M, Brillet PY, Fekih ZE, Bruno RM, Bihan H, Cosson E. Epicardial adipose tissue volume and arterial stiffness in people living with diabetes: the METAB-CV-PWV study. Cardiovasc Diabetol. 2025 Oct 15;24(1):400. doi: 10.1186/s12933-025-02933-z. PMID 41094476